CLINICAL TRIAL: NCT00951223
Title: Observational Prospective Registry of the Efficacy, Safety, and Adherence to Therapy of Infergen® (Interferon Alfacon 1) in Patients Chronically Infected With Hepatitis C Virus
Brief Title: Observational Prospective Registry of the Efficacy, Safety, and Adherence to Infergen® in Patients Infected With Hep C
Acronym: REACHSVR
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Enrollment
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CIFN 003
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — interferon alfacon-1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Chronic Hepatitis C: HCV positive patients who have failed previous HCV therapy This observational prospective registry is designed to evaluate the safety, adherence, and efficacy of prescribed, patientadministered therapy with Infergen® (Interferon alfacon-1) and other prescribed therapies in patients chronically infected with HCV. The primary endpoint for efficacy will be the SVR rate at 24 weeks after therapy ends. Safety will be assessed by monitoring AEs, reduction/discontinuation of therapy because of AEs, routine laboratory results and by other means determined by the Investigator
  Interventions: Drug: Infergen® (Interferon alfacon-1)

INTERVENTIONS:
Drug: Infergen® (Interferon alfacon-1) — Infergen at either the 15 mcg or 9 mcg dose given per Providers instructions, with or without weight based ribavirin
  Other Names: INF

SUMMARY:
This observational prospective registry is designed to evaluate the safety, adherence, and efficacy of prescribed, patient-administered therapy with Infergen® (Interferon alfacon 1) and other prescribed therapies in patients chronically infected with HCV. The primary endpoint for efficacy will be the SVR rate at 24 weeks after therapy ends.

DETAILED DESCRIPTION:
This registry plans to enroll 1000 patients at 75 clinical sites across the United States.

Potentially eligible patients will be anti-HCV antibody-positive and have detectable serum or plasma HCV RNA. Patients can have any HCV genotype; they also can be antiviral treatment-naïve or have a history of either nonresponse or relapse to previous antiviral therapy. Patients can roll over directly from current interferon (IFN) therapy into registry Infergen therapy, but the average washout period will be <1 month. Rollovers will occur after 4, 12, or 24 weeks of IFN therapy. Patients coinfected with HBV or HIV can be included in the registry.

Each investigator participating in this registry will employ his or her discretion and standard clinical practice to determine when to see the patient in the clinic, how to manage the patient's drug regimen, and how best to monitor the patient's response and tolerance to therapy.The decision to enroll a patient and start therapy with Infergen and other prescribed therapies may be guided by historic biopsy results, or the patient can undergo liver biopsy at the investigator's discretion. Biopsy is not a prerequisite, however, if the investigator believes it to be unnecessary. When a patient's treatment is expected to require significant dose modification and/or more intensive monitoring because of comorbid conditions, enrolling the patient in the registry is at the investigator's discretion. For purposes of the registry, data will be collected at baseline; at Weeks 4, 12, 24, and 48 from the start of therapy; and at follow-up visits 4 and 24 weeks after treatment ends.

Safety will be assessed by monitoring AEs, reduction/discontinuation of therapy because of AEs, routine laboratory results and by other means determined by the investigator. Adherence over the course of therapy will also be evaluated, taking into account physician-directed dose reduction or cessation, patients' self-reports of compliance, and the return of used and unused medication to each scheduled visit.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to consent to data being collected and provided to the Duke Clinical Research Institute (DCRI) and Three Rivers Pharmaceuticals
2. Able and willing to give written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization, and to comply with the requirements of the registry protocol
3. Anti-HCV antibody-positive
4. HCV RNA concentration >100,000 IU/mL on reverse transcriptase-polymerase chain reaction (RT-PCR) assay at baseline or >90 days before the baseline visit
5. Deemed by the investigator to be an appropriate patient for treatment with Infergen and other prescribed medications
6. Baseline CD4 count >200 cells/mm3 (human immunodeficiency virus [HIV]-HCV coinfected patients)
7. Women: must be documented to be surgically sterile, be postmenopausal (defined as >2 years without menses), or agree to use 2 forms of effective contraception during the registry and for 6 months after receiving the final dose of study drug. Men: must agree to use 2 forms of effective contraception during the registry and for 6 months after receiving the final dose of study drug, and their partners of childbearing potential must not be pregnant at screening.
8. Women: must not be lactating and, if of childbearing potential, must have a negative serum pregnancy test result at the baseline visit
9. Age >18 years

Exclusion Criteria:

1. Unable to complete all clinic visits and comply with registry procedures, including self-injection of Infergen
2. Known hypersensitivity to alpha-interferons or any component of the product
3. Decompensated hepatic disease
4. Autoimmune hepatitis
5. Hemoglobinopathies (i.e., thalassemia or sickle cell anemia)
6. Any other condition that, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in and completing the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Community Gastrointestinal Practices as well as Academic Centers will be asked to participate
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Determine the incidence of SVR, defined as undetectable HCV RNA measured 24 weeks after therapy ends, associated with prescribed, patient-administered therapy with Infergen® (Interferon alfacon 1) in patients chronically infected with HCV. | 24 weeks post end of therapy

SECONDARY OUTCOMES:
Capture of defined adverse events (AEs),dose changes or cessation, and adherence to the prescribed dose of Infergen and other prescribed therapies over the course of treatment | Treatment weeks 4, 12, 24, 48, and Follow-Up weeks 4 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Muir, MD, Principal Investigator — DCRI